CLINICAL TRIAL: NCT05409703
Title: The Effect of Reiki on Executive Nurses on Psychological Empowerment, Happiness, Emotion Management and Work Engagement
Brief Title: The Effect of Reiki on Executive Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zehra Bayram (Other)
Responsible Party: Sponsor-Investigator, Zehra Bayram, Nurse, Cukurova University
Organization: Cukurova University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 92372714
Record Dates: First submitted 2022-05-27; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Reiki Therapy
Keywords: Executive Nurses; Reiki; Psychological Empowerment; Happiness; Emotion Management
MeSH Terms: interventions — Therapeutic Touch

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental study.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effect of Reiki on Executive Nurses on Psychological Empowerment, Happiness (Experimental): Reiki application will take 45 minutes.
  Interventions: Behavioral: reiki therapy
- The Effect of Reiki on Executive Nurses on Emotion Management and Work Engagement (No Intervention): No treatment was applied to the patients in the control group other than their routine care.

INTERVENTIONS:
Behavioral: reiki therapy — reiki therapy for nurses
  Arms: The Effect of Reiki on Executive Nurses on Psychological Empowerment, Happiness

SUMMARY:
In this study, the traditional Usui Reiki protocol was applied for distant healing. Each session; It was applied approximately once a week, for 30 minutes, for two weeks. A certified Reiki practitioner (one of the researchers) received an energy transfer from his home, 80 km away. The practitioner is trained in the reiki line and has been practicing and continuing to practice reiki for over 5 years.

DETAILED DESCRIPTION:
The practitioner made an appointment over the phone to conduct individual sessions during the morning hours when each participant was available. Before the first session, the online pre-assessment tools (Google form) of the study were delivered to the participant, and then a statement of intent was sent to the participant. The person who will take the session is requested to be in a comfortable position. During the application, he/she can talk, sleep, work if he/she wishes. However, he was warned not to use tools and cutting tools. The second session will be held at the same time, one week later, and the online final evaluation forms were asked to be filled one day later. The group will be re-evaluated after 21 days. No intervention was made in the control group. The same measurement tools were used in all groups.

ELIGIBILITY:
Inclusion Criteria:

Holding a managerial position, Executive nurses who have not received reiki therapy before will be included in the study.

Exclusion Criteria:

Previous or current reiki therapy Reiki practitioner or instructor, Nurses who are not in a managerial position will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
The Effect of Reiki on Executive Nurses on Psychological Empowerment | Scales are filled after 6 weeks of application.
  Emotion Management Skills Scale The "Emotion Management Skills Scale" (DYLL) developed by Çeçen (2006) consists of 8 positive (2, 8, 10, 12, 17, 19, 21, 26), 20 negative (1, 3, 4, 5 , 6, 7, 9, 11, 13, 14, 15, 16, 18, 20, 22, 23, 24, 25, 27, 28) consists of 28 items and 5 sub-dimensions.The highest score that can be obtained from the scale is 140, and the lowest score is 28. High scores indicate that the individual is competent in managing his emotions. The Cronbach Alpha internal reliability coefficient of the Emotion management skills scale developed by Çeçen (2006) is 0.83.
The Effect of Reiki on Executive Nurses on Emotion Management and Work Engagement | Scales are filled after 6 weeks of application.
  Oxford Happiness Scale The Oxford Happiness Scale Short Form (OMÖ-K) was developed by Hills and Argyle (2002), and adapted into Turkish by Doğan and Akıncı-Çötok (2011). In the adaptation study, the internal consistency coefficient was calculated as .75 and the test-retest reliability coefficient as .87. The scale consists of 7 items and is a 5-point Likert type scale. High scores from the scale indicate a high level of happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Kuşçu Karatepe, phD, Principal Investigator — Osmaniye Korkut Ata University
Locations (1):
- Zehra Bayram, Osmaniye, Turkey (Türkiye)